CLINICAL TRIAL: NCT00637481
Title: A Phase I Prevention Study of Atorvastatin in Women at Increased Risk for Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NCI-2009-00859; NCI-2009-00859 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000653466; 2006-0185 (Other: M D Anderson Cancer Center); MDA05-6-01 (Other: DCP); N01CN35159 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2008-03-17; First posted 2008-03-18 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Atypical Ductal Breast Hyperplasia; Breast Cancer; Ductal Breast Carcinoma in Situ; Lobular Breast Carcinoma in Situ
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Neoplasms; Breast Carcinoma In Situ | interventions — Atorvastatin

ARMS (4):
- Arm I (lower dose atorvastatin calcium) (Experimental): Participants receive oral atorvastatin once daily for 3 months.
  Interventions: Drug: atorvastatin calcium; Other: laboratory biomarker analysis
- Arm II (atorvastatin calcium) (Experimental): Participants receive oral atorvastatin (at a higher dose than in arm I) once daily for 3 months.
  Interventions: Drug: atorvastatin calcium; Other: laboratory biomarker analysis
- Arm III (higher dose atorvastatin calcium) (Experimental): Participants receive oral atorvastatin (at a higher dose than in arm II) once daily for 3 months.
  Interventions: Drug: atorvastatin calcium; Other: laboratory biomarker analysis
- Arm IV (no intervention) (Other): Participants do not receive treatment. Participants undergo blood sample collection and fine needle aspiration of breast tissue at baseline and at 3 months for correlative biomarker studies.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: atorvastatin calcium — Given orally
  Other Names: CI-981; Lipitor
  Arms: Arm I (lower dose atorvastatin calcium); Arm II (atorvastatin calcium); Arm III (higher dose atorvastatin calcium)
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Chemoprevention is the use of certain drugs to keep cancer from forming. The use of atorvastatin (Lipitor) may prevent breast cancer. This randomized phase I trial is studying the best dose of atorvastatin in preventing breast cancer in women at increased risk for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the minimum biological effective dose (MBED) of atorvastatin required to induce modulation in the proliferation marker, Ki-67, in breast tissue of women who are at high risk to develop breast cancer. We will evaluate pre- and post atorvastatin treatment (4 dose levels) expression of Ki-67 in samples obtained via FNA from breast tissue of women at high risk for breast cancer. This specific aim tests the hypothesis that treatment with atorvastatin will induce a decrease in Ki-67.

SECONDARY OBJECTIVES:

I. To evaluate atorvastatin induced modulation of breast cancer biomarkers markers (EGFR, P-EGFR, ER, p21, p27, bcl-2, CC3, cytology) and drug related markers (LXR, total cholesterol, LDL, HDL, CRP) in women who are at high risk to develop breast cancer.

II. To determine plasma and tissue levels of atorvastatin and two of its hydroxylated metabolites (ohydroxyatorvastatin and p-hydroxyatorvastatin) in women who are treated with atorvastatin and to correlate these levels with Ki-67 levels. III. To correlate changes in Ki-67 and the above-described panel of biomarkers with HMG-CoA reductase genotype.

OUTLINE: Participants are randomized to 1 of 4 arms.

ARM I: Participants receive oral atorvastatin once daily for 3 months.

ARM II: Participants receive oral atorvastatin (at a higher dose than in arm I) once daily for 3 months.

ARM III: Participants receive oral atorvastatin (at a higher dose than in arm II) once daily for 3 months.

ARM IV: Participants do not receive treatment. Participants undergo blood sample collection and fine needle aspiration of breast tissue at baseline and at 3 months for correlative biomarker studies.

ELIGIBILITY:
Inclusion Criteria:

* Women at increased risk for breast cancer, defined by one of the following:

  * 5 year projected Gail risk of greater than 1.67%
  * Previous diagnosis of atypical hyperplasia (AH) or lobular carcinoma in situ (LCIS) (per participating institution's pathology review), or ductal carcinoma in situ (participants could have received any type of surgery and radiation as long as they have an intact opposite breast)
* The participant must have been properly informed of the study and must sign an informed consent to be able to be enrolled in the study; the informed consent document must be signed, witnessed, and dated prior to start of the study
* Normal physical exam and bilateral mammogram that shows no evidence of suspicious, malignant disease, or uncharacterized lesions within last 12 months and no evidence of any active other cancer
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky greater than or equal to 70%)
* Leukocytes greater than 3,000/uL
* Platelets greater than 100,000/uL
* Total bilirubin within normal institutional limits
* AST (SGOT)or /ALT (SGPT) =< 1.5 X institutional ULN
* Creatinine within normal institutional limits
* CPK, PTT, PT within normal institutional limits (up to 1 month prior to randomization)
* The effects of atorvastatin on the developing human fetus at the recommended therapeutic dose are unknown; for this reason, women of child-bearing potential must agree to use adequate contraception (barrier method of birth control (IUD); abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her study physician immediately

Exclusion Criteria:

* Any type of active invasive cancer
* Bilateral mastectomy
* Use of oral contraceptives; androgens; luteinizing-hormone-releasing-hormone (LHRH) analogs, prolactin inhibitors, antiandrogens, tamoxifen, raloxifen, or aromatase inhibitors; women who discontinue these drugs at least 3 months prior to study enrollment will be eligible
* Chronic medical condition that requires regular use of statins or steroids (unless participants have discontinued these drugs 1 month prior to enrollment)
* Participants may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to atorvastatin
* Psychiatric condition, including history of clinical depression, or addictive disorder that would preclude obtaining informed consent or would interfere with compliance; uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because atorvastatin is a Class X agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with atorvastatin breast feeding should be discontinued if the mother is treated with atorvastatin

Ages: 18 Years to 72 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2008-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Atorvastatin induced changes in proliferation rate measured by Ki-67 | Baseline to 3 months
  A single proliferation rate at each time period is calculated for each participant based on the proportion cells expressing KI-67.

SECONDARY OUTCOMES:
Cytologic evaluation of FNA samples | Baseline
Cytologic evaluation of FNA samples | 3 months
Proliferation and apoptosis analysis of FNA samples | Baseline
Proliferation and apoptosis analysis of FNA samples | 3 months
Inflammatory and lipid profile markers | Up to 3 months
Genotypic analysis | Baseline
Measurement of atorvastatin and its metabolites in serum and breast tissue | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States